CLINICAL TRIAL: NCT02774980
Title: Cognitive Markers of Response to Treatment in Resistant Depression
Acronym: DEP-ICOR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 14-AOI-07
Record Dates: First submitted 2016-05-03; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Recurrent depression

SUMMARY:
Patients with depression are frequently treatment resistant. Clinical manifestations of depression are various, but cognitive dysfunctions are commonly present. Many factors are involved in treatment resistance. As no biological marker is available, clinical markers could be considered in predicting response to antidepressive treatment.

The aim of this study is to investigate the relation between the cognitive changes and the remission of depressive symptoms in patients with recurrent depression (Stage 2 of Thase and Rush classification).

To explore the dynamics of cognitive dimension associated to clinical and functional remission, the investigators will observe neurocognitive functioning before and after introducing a new antidepressive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be aged from 40 to 70, with a major depressive episode diagnosis with a 2 stage degree of resistance.

Exclusion Criteria:

* Patients with major depressive episode during more of 12 months
* Alzheimer dementia or related disease (CIM 10)
* Score Hamilton Depression Rating Scale (HDRS) < 18

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a major depressive episode diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Clinic assessments: Score BDI - II | Change from the baseline score BDI-II at 12 months after introducing the new therapy
  The investigators will conduct clinical assessments. A baseline will be drawn in the acute phase (V1) before modifying the antidepressive therapy; 2 weeks after treatment change, patient will be clinically assessed by his psychiatrist. A complete assessment will be done 6 months and 12 months after introducing the new therapy.
Functional assessments : Score Sheehan Disability Scale (SDS) | Change from the baseline Score Sheehan Disability Scale (SDS) at 12 months after introducing the new therapy
  The investigators will conduct functional assessments. A baseline will be drawn in the acute phase (V1) before modifying the antidepressive therapy; 2 weeks after treatment change, patient will be functional assessed by his psychiatrist. A complete assessment will be done 6 months and 12 months after introducing the new therapy.
Neuropsychologic assessments: M.M.S.E. (Mini Mental Score Evaluation) | Change from the baseline Score M.M.S.E. (Mini Mental Score Evaluation) at 12 months after introducing the new therapy
  The investigators will conduct neuropsychologic assessments. A baseline will be drawn in the acute phase (V1) before modifying the antidepressive therapy; A complete assessment will be done 6 months and 12 months after introducing the new therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nelly Darmon, Principal Investigator — CHU of Nice
Locations (1):
- Hopital Pasteur, Nice, France

IPD SHARING:
Plan to Share IPD: No